CLINICAL TRIAL: NCT04283981
Title: Comparison of Operating Room Time Length With the Use of Virtual Surgical Planning Versus Conventional Treatment of Mandible Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Principal Investigator, Simon Young, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-19-1074
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Device: Control group without use of VSP
- Treatment Group (Experimental)
  Interventions: Device: Treatment Group with use of VSP

INTERVENTIONS:
Device: Control group without use of VSP — The control group will include patients that undergo mandibular reconstruction via open reduction internal fixation (intraoral or extraoral approach) in standard fashion (without virtual surgical planning assistance and occlusal splint)
  Arms: Control Group
Device: Treatment Group with use of VSP — The treatment group corresponds to patients undergoing mandibular reconstruction via open reduction internal fixation (intraoral or extraoral approach) utilizing virtual surgical planning via 3D Systems, bite registration and fabrication of occlusal splint via intraoral digital scanner, and mandibular hardware
  Arms: Treatment Group

SUMMARY:
The purpose of this trial is to compare operating room time between conventional treatment techniques [without Virtual surgical Planning (VSP)] versus treatment with use of Virtual surgical Planning (VSP) in patients that undergo mandibular reconstruction via open reduction internal fixation (ORIF).

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Complex mandible fracture (at least two fractures) that require ORIF of at least one fracture. This will exclude condylar fractures

Exclusion Criteria:

* Patient refusal to participate in study
* Infected mandible fracture
* Closed reduction treatment of mandible fracture
* Fractures older than 2-3 weeks at the time of treatment
* Other concomitant mid-facial bone fractures (ie, zygomaticomaxillary complex (ZMC), Lefort fractures)
* Other etiologies than trauma of the mandibular fracture or pathologic fracture secondary to benign or malignant pathology that may require resection
* Pregnant patients will NOT be excluded from the study
* Co-morbidities (auto-immune disease, osteoporosis, titanium or metal allergy, uncontrolled diabetes (A1c greater than 8)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Woernley, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 15 | 13
Completed | 9 | 7
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.3) | 26.7 (8.5) | 30.75 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 6 | 7 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16
Mandible Fracture Severity as Assessed by the Mandible Injury Severity Score [Mean (Standard Deviation); unit: score on a scale] — Mandible Injury Severity Score assess the severity of mandibular fractures. The total score ranges from 5 to 52, a higher score indicating a worse outcome
  score on a scale | 15.7 (9.4) | 18.3 (8) | 16.8 (8.8)
Number of Mandible Fractures [Mean (Standard Deviation); unit: fractures] | 2.33 (.50) | 2.13 (.38) | 2.24 (.45)

OUTCOME MEASURES:

1. Primary Outcome: The Time Taken to Complete an Open Reduction Internal Fixation (ORIF)
Description: The time taken to complete an Open Reduction Internal Fixation (ORIF) [referred to as the "plating time"] was defined as beginning after dissection was complete and fractures were initially reduced, and ending after all fracture sites were fixated with the final screw placed.
Time Frame: from start of ORIF to end of ORIF (about 2-3 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
minutes | 54.6 (28.9) | 34 (12.5)

2. Secondary Outcome: Number of Participants With Malocclusion
Time Frame: 1 week after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Malocclusion
Time Frame: 3 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With Malocclusion
Time Frame: 6 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 2 | 0

5. Secondary Outcome: Number of Participants With Fractures That Are Not Well Aligned
Time Frame: 1 week after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Fractures That Are Not Well Aligned
Time Frame: 3 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Fractures That Are Not Well Aligned
Time Frame: 6 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Infections
Time Frame: 1 week after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 1 | 1

9. Secondary Outcome: Number of Participants With Infections
Time Frame: 3 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Infections
Time Frame: 6 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

11. Secondary Outcome: Type of Archbars Used in ORIF
Description: Archbars are used for fixating jaws during the treatment of mandible fractures. Archbars are anchored onto both jaws (that is, onto the maxillar/upper jaw, and onto the mandibular/lower jaw); therefore, each participant receives 2 arch bars, one for each jaw. Data are reported categorically as the type of arch bar received for a jaw.
Time Frame: from start of ORIF to end of ORIF (about 2-3 hours)
Measure: Number; unit: archbars
Units Other Than Participants: jaws
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Number analyzed (jaws) | 18 | 14
archbars
  None | 2 | 0
  Erich | 10 | 9
  Biomet Omnimax | 2 | 0
  Stryker SMARTLock Hybrid | 0 | 2
  Synthes MatrixWAVE | 4 | 1
  Ivy Loops | 0 | 2

12. Secondary Outcome: Number of Participants Whose Occlusal Splint Fit Appropriately
Time Frame: from start of ORIF to end of ORIF (about 2-3 hours)
Population: Data were not collected for 9 participants in the control group
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 7 | 0
Participants | 7 |

13. Secondary Outcome: Type of Surgical Approach to the Fracture Site
Description: The type of surgical approach to the fracture site is reported categorically as either extraoral or intraoral. This is counted based on each fracture approached surgically (a participant may have more than 1 approach if they had more than 1 fracture site).
Time Frame: from start of ORIF to end of ORIF (about 2-3 hours)
Measure: Number; unit: specified approaches
Units Other Than Participants: fracture sites
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Number analyzed (fracture sites) | 14 | 12
specified approaches
  Intraoral | 7 | 5
  Extraoral | 7 | 7

14. Secondary Outcome: Number of Participants Who Required Intraoperative Surgical Revisions
Time Frame: from start of ORIF to end of ORIF (about 2-3 hours)
Population: Data were not collected for 9 participants in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 7
Participants |  | 0

15. Secondary Outcome: Distance of Maximal Interincisal Opening
Description: Maximal interincisal opening is the maximum distance a person can open their mouth between their upper and lower incisors measured in millimeters.
Time Frame: 6 weeks after ORIF
Population: Data were not collected for 4 participants in the control group. Data were not collected for 3 participants in the treatment group.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 5 | 4
millimeters | 34.6 (8.16) | 31.8 (6.83)

16. Secondary Outcome: Number of Participants With Hardware Failure
Description: Number of Participants with hardware failure as defined as plate fracture or screw loosening
Time Frame: from baseline to 6 weeks after ORIF
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post-surgery
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/13
Other Adverse Events (participants affected / at risk) | 2/15 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=15) | Treatment Group (N=13)
Postoperative Infection (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=15) | Treatment Group (N=13)
Post-operative Malocclusion of Teeth (Surgical and medical procedures) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04283981/Prot_SAP_000.pdf